CLINICAL TRIAL: NCT02494934
Title: A Randomized Comparison of Individual Cognitive-behavioural Therapy and Pelvic Floor Rehabilitation in the Treatment of Provoked Vestibulodynia
Brief Title: Effectiveness of Cognitive Behavioural Therapy and Physical Therapy for Provoked Vestibulodynia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Caroline Pukall, Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 379631
Record Dates: First submitted 2015-06-30; First posted 2015-07-10 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Vulvar Vestibulitis
MeSH Terms: conditions — Vulvar Vestibulitis | interventions — Cognitive Behavioral Therapy; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive-behavioural therapy (Experimental): Eight sessions of psychotherapy incorporating cognitive-behavioural and sex therapy interventions.
  Interventions: Behavioral: cognitive-behavioural therapy
- physical therapy (Experimental): Eight sessions of physical therapy targeting the pelvic floor muscles.
  Interventions: Behavioral: physical therapy

INTERVENTIONS:
Behavioral: cognitive-behavioural therapy — The CBT program was adapted from a previously used group CBT program and included the following procedures: (1) education about PVD; (2) collaborative re-conceptualization of PVD as a multi-factorial pain condition; (3) desensitization exercises; (4) diaphragmatic breathing and other relaxation techniques; (5) discussion about and techniques for increasing sexual desire and arousal; (6) sexual communication skills training; (7) instructions on carrying out PFM exercises; (8) instructions on the use of silicone vaginal dilators to do progressive vaginal penetration activities at home; and (9) informal and formal cognitive restructuring techniques and the use of coping self-statements.
  Arms: Cognitive-behavioural therapy
Behavioral: physical therapy — The PT treatment protocol included the following procedures: (1) education about PVD; (2) targeted PFM exercises focused on contraction and relaxation including in-session practice and feedback; (3) manual techniques; (4) surface electromyographic biofeedback (sEMG); (5) progressive vaginal penetration activities through the use of four silicone vaginal dilators of varied diameter; (6) stretches of the hip muscles; (7) deep breathing and global body relaxation exercises; and (8) additional methods of managing pain and counseling about different sexual positions.
  Arms: physical therapy

SUMMARY:
The purpose of the study was to compare the effectiveness of cognitive behavioural therapy (CBT) and physical therapy (PT) on pain and psychosexual outcomes in women with provoked vestibulodynia (PVD).

DETAILED DESCRIPTION:
Provoked vestibulodynia (PVD) is the most common condition leading to painful intercourse and is currently best understood within a biopsychosocial framework. Although the usefulness of non-medical treatment options for vulvar pain is recognized by many, there is limited research investigating the effectiveness of these treatments using a biopsychosocial approach to outcome measurement. Furthermore, there is little evidence to support the mechanisms by which these treatments lead to pain reduction. This study aimed to address these gaps by investigating two non-medical treatment options: individual cognitive-behavioural therapy (CBT) and physical therapy (PT).

ELIGIBILITY:
Inclusion Criteria:

* fluent in English
* vulvar pain with attempted vaginal penetration for at least 6 months
* pain limited to vulvar vestibule during cotton swab test

Exclusion Criteria:

* other serious medical, psychiatric, or other pain conditions
* generalized vulvodynia and/or significant vaginismus (i.e., not able to have at least one finger inserted vaginally)
* current pregnancy, breastfeeding, or being less than 6 months postpartum
* unwillingness to abstain from other treatments for their PVD pain during the course of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
change from baseline in pain with sexual intercourse at 12 weeks | Baseline, 12 weeks
  measured on an 11-point numerical rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Pukall, PhD, Principal Investigator — Queen's University